CLINICAL TRIAL: NCT02928198
Title: Bifurcation ABSORB OCT Trial
Acronym: BISORB OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: J.J. Wykrzykowska (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, J.J. Wykrzykowska, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL50172.018.14
Record Dates: First submitted 2016-09-09; First posted 2016-10-10 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Ischemia; Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Coronary Bifurcation Lesions; Arterial Occlusive Lesions; Infarction; Myocardial Infarction; Arteriosclerosis
Keywords: Tomography, Optical Coherence; Percutaneous Coronary Intervention; Cardiac Catheterization; Coronary Biovascular Scaffold
MeSH Terms: conditions — Myocardial Ischemia; Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Infarction; Myocardial Infarction; Arteriosclerosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Fenestration (Active Comparator): Fenestration of the Absorb Biovascular Scaffold towards the side-branch
  Interventions: Device: ABSORB BVS
- No Fenestration (Active Comparator): No fenestration of the Absorb Biovascular Scaffold towards the side-branch
  Interventions: Device: ABSORB BVS

INTERVENTIONS:
Device: ABSORB BVS

SUMMARY:
The Bifurcation ABSORB OCT Trial is a prospective, randomized (1:1) evaluation of the efficacy and performance of single ABSORB everolimus eluting bioresorbable vascular scaffold provisional strategy in the treatment of (a) coronary bifurcation lesion(s) in consecutive subjects with and without fenestration towards the side branch.

Patients included in this study will be divided into three different cohorts:

* Cohort A (patient 1-20): Angiographic FU with OCT at 12 months.
* Cohort B (patient 21-40): Angiographic FU with OCT at 24 months.
* Cohort C (patient 41-60): Angiographic FU with OCT at 36 months.

All patients will also have telephone FU at 30 days, 12, 24 and 36 months.

Inclusion of patients in the BISORB OCT trial stopped in November 2016 after safety concerns of the ABSORB BVS were reported. BISORB OCT included 3 patients, which were all included in the Academic Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Subject has a bifurcation lesion involving a side-branch larger than 2 mm and having main branch involvement (Medina 0,0,1 lesions are excluded).
* Subject must agree to undergo all clinical investigation plan-required follow-up visits and to undergo follow-up angiography and optical coherence tomography.
* Subject is able to verbally confirm understanding and he/she or his/her legally authorized representative provides written informed consent prior to any Clinical Investigation related procedure,as approved by the appropriate Ethics Committee.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is presenting with a STEMI
* Subject has a true bifurcation lesion where a priori two scaffold/stent strategy is planned.
* Subject has known hypersensitivity or contraindication to contrast, aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel, prasugrel and ticagrelor, inclusive), everolimus, poly (L-lactide), poly (DL-lactide), cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
* Known renal insufficiency (eg. estimated Glomerular Filtration Rate (eGFR) <60mL/min/1.73m2 or serum creatinine level of >2.5mg/dL or subject on dialysis)
* Subject with a limited life expectancy less than one year.
* Subject is belonging to a vulnerable population (per investigator's judgment, e.g., subordinate hospital staff) or subject unable to read or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number and appearance of jailed side branch struts, as assessed with three-dimensional OCT - Cohort A | 12 months
  3D reconstruction assessment is done visually and the number of strut free compartments are categorized as follows: Non-jailed side branch or jailed side branch. Non-jailed side branch is defined as either no strut over the sidebranch is present or 1 of the BVS struts is present over the side branch but does not compartmentalize the side branch. Jailed side branch is defined as the BVS struts separate the side branch ostium into n compartments. The distribution of the struts creates different patterns of compartments: V, T, H, double V, double T, and double H.

SECONDARY OUTCOMES:
Number and appearance of jailed side branch struts, as assessed with three-dimensional OCT - All cohorts | Baseline
  3D reconstruction assessment is done visually and the number of strut free compartments are categorized as follows: Non-jailed side branch or jailed side branch. Non-jailed side branch is defined as either no strut over the sidebranch is present or 1 of the BVS struts is present over the side branch but does not compartmentalize the side branch. Jailed side branch is defined as the BVS struts separate the side branch ostium into n compartments. The distribution of the struts creates different patterns of compartments: V, T, H, double V, double T, and double H.
Number and appearance of jailed side branch struts, as assessed with three-dimensional OCT - Cohort B | 24 months
  3D reconstruction assessment is done visually and the number of strut free compartments are categorized as follows: Non-jailed side branch or jailed side branch. Non-jailed side branch is defined as either no strut over the sidebranch is present or 1 of the BVS struts is present over the side branch but does not compartmentalize the side branch. Jailed side branch is defined as the BVS struts separate the side branch ostium into n compartments. The distribution of the struts creates different patterns of compartments: V, T, H, double V, double T, and double H.
Number and appearance of jailed side branch struts, as assessed with three-dimensional OCT - Cohort C | 36 months
  3D reconstruction assessment is done visually and the number of strut free compartments are categorized as follows: Non-jailed side branch or jailed side branch. Non-jailed side branch is defined as either no strut over the sidebranch is present or 1 of the BVS struts is present over the side branch but does not compartmentalize the side branch. Jailed side branch is defined as the BVS struts separate the side branch ostium into n compartments. The distribution of the struts creates different patterns of compartments: V, T, H, double V, double T, and double H.
Incomplete strut apposition in the bifurcation region - All cohorts | Baseline
  Present when, in case of an ABSORB BVS, the abluminal surface of the polymeric strut (black box) is separated from the vessel wall by flush, between 0.5mm proximal and 0.5mm distal of the side branch.
Incomplete strut apposition in the bifurcation region - Cohort A | 12 months
  Present when, in case of an ABSORB BVS, the abluminal surface of the polymeric strut (black box) is separated from the vessel wall by flush, between 0.5mm proximal and 0.5mm distal of the side branch.
Incomplete strut apposition in the bifurcation region - Cohort B | 24 months
  Present when, in case of an ABSORB BVS, the abluminal surface of the polymeric strut (black box) is separated from the vessel wall by flush, between 0.5mm proximal and 0.5mm distal of the side branch.
Incomplete strut apposition in the bifurcation region - Cohort C | 36 months
  Present when, in case of an ABSORB BVS, the abluminal surface of the polymeric strut (black box) is separated from the vessel wall by flush, between 0.5mm proximal and 0.5mm distal of the side branch.
Number of embedded and protruded ABSORB BVS struts per region - All cohorts | Baseline
  Embedded struts are defined as present when more than one-half thickness of the strut was impacted into the vessel wall.
Number of embedded and protruded ABSORB BVS struts per region - Cohort A | 12 months
  Embedded struts are defined as present when more than one-half thickness of the strut was impacted into the vessel wall.
Number of embedded and protruded ABSORB BVS struts per region - Cohort B | 24 months
  Embedded struts are defined as present when more than one-half thickness of the strut was impacted into the vessel wall.
Number of embedded and protruded ABSORB BVS struts per region - Cohort C | 36 months
  Embedded struts are defined as present when more than one-half thickness of the strut was impacted into the vessel wall.
Incomplete strut coverage in the bifurcation region - Cohort A | 12 months
  Absence of strut coverage at the side-branch ostium is defined when one of the strut corners preserved a right angle shape without signs of neointimal tissue, between 0.5mm proximal and 0.5mm distal of the side branch.
Incomplete strut coverage in the bifurcation region - Cohort B | 24 months
  Absence of strut coverage at the side-branch ostium is defined when one of the strut corners preserved a right angle shape without signs of neointimal tissue, between 0.5mm proximal and 0.5mm distal of the side branch.
Incomplete strut coverage in the bifurcation region - Cohort C | 36 months
  Absence of strut coverage at the side-branch ostium is defined when one of the strut corners preserved a right angle shape without signs of neointimal tissue, between 0.5mm proximal and 0.5mm distal of the side branch.
The number of non-apposed side branch (NASB) struts - All cohorts | Baseline
  Non-apposed side branch struts are defined as struts overlying the ostium of a sidebranch, post-scaffold deployment and at follow up.
The number of non-apposed side branch (NASB) struts - Cohort A | 12 months
  Non-apposed side branch struts are defined as struts overlying the ostium of a sidebranch, post-scaffold deployment and at follow up.
The number of non-apposed side branch (NASB) struts - Cohort B | 24 months
  Non-apposed side branch struts are defined as struts overlying the ostium of a sidebranch, post-scaffold deployment and at follow up.
The number of non-apposed side branch (NASB) struts - Cohort C | 36 months
  Non-apposed side branch struts are defined as struts overlying the ostium of a sidebranch, post-scaffold deployment and at follow up.
Tissue in-between non-apposed side branch (NASB) struts - Cohort A | 12 months
  Tissue in-between NASB struts is defined as any tissue between two NASB ABSORB struts more than two times the polymer thickness.
Tissue in-between non-apposed side branch (NASB) struts - Cohort B | 24 months
  Tissue in-between NASB struts is defined as any tissue between two NASB ABSORB struts more than two times the polymer thickness.
Tissue in-between non-apposed side branch (NASB) struts - Cohort C | 36 months
  Tissue in-between NASB struts is defined as any tissue between two NASB ABSORB struts more than two times the polymer thickness.
Mean/Minimal Lumen diameter/area - All cohorts | Baseline
  Lumen diameter and lumen area are measured at the (neo-)intima layer of the vessel wall, both pre- and post-scaffold deployment and at follow up. At baseline this is usually outside the scaffold diameter/area and at follow up into the scaffold diameter/area
Mean/Minimal Lumen diameter/area - Cohort A | 12 months
  Lumen diameter and lumen area are measured at the (neo-)intima layer of the vessel wall, both pre- and post-scaffold deployment and at follow up. At baseline this is usually outside the scaffold diameter/area and at follow up into the scaffold diameter/area
Mean/Minimal Lumen diameter/area - Cohort B | 24 months
  Lumen diameter and lumen area are measured at the (neo-)intima layer of the vessel wall, both pre- and post-scaffold deployment and at follow up. At baseline this is usually outside the scaffold diameter/area and at follow up into the scaffold diameter/area
Mean/Minimal Lumen diameter/area - Cohort C | 36 months
  Lumen diameter and lumen area are measured at the (neo-)intima layer of the vessel wall, both pre- and post-scaffold deployment and at follow up. At baseline this is usually outside the scaffold diameter/area and at follow up into the scaffold diameter/area
Mean/Minimal Scaffold diameter/area - All cohorts | Baseline
  Scaffold diameter and scaffold area are measured at the abluminal border of the polymeric struts (black boxes), both post-scaffold deployment and at follow up.
Mean/Minimal Scaffold diameter/area - Cohort A | 12 months
  Scaffold diameter and scaffold area are measured at the abluminal border of the polymeric struts (black boxes), both post-scaffold deployment and at follow up.
Mean/Minimal Scaffold diameter/area - Cohort B | 24 months
  Scaffold diameter and scaffold area are measured at the abluminal border of the polymeric struts (black boxes), both post-scaffold deployment and at follow up.
Mean/Minimal Scaffold diameter/area - Cohort C | 36 months
  Scaffold diameter and scaffold area are measured at the abluminal border of the polymeric struts (black boxes), both post-scaffold deployment and at follow up.
Neointima thickness - Cohort A | 12 months
  Neointima thickness of the ABSORB BVS is measured from the endoluminal border of the black box to the lumen contour.
Neointima thickness - Cohort B | 24 months
  Neointima thickness of the ABSORB BVS is measured from the endoluminal border of the black box to the lumen contour.
Neointima thickness - Cohort C | 36 months
  Neointima thickness of the ABSORB BVS is measured from the endoluminal border of the black box to the lumen contour.
Scaffold pattern irregularities - All cohorts | Baseline
  Scaffold pattern irregularities are defined when struts are found in locations incongruent with the scaffold pattern, this is measured post-scaffold deployment and at follow up. They are classified into 2 categories: 1) 2 struts overhanging each other in the same angular sector of the lumen perimeter, with or without malapposition; and/or 2) isolated struts located more or less at the center of the vessel without obvious connection to the expected adjacent strut pattern.
Scaffold pattern irregularities - Cohort A | 12 months
  Scaffold pattern irregularities are defined when struts are found in locations incongruent with the scaffold pattern, this is measured post-scaffold deployment and at follow up. They are classified into 2 categories: 1) 2 struts overhanging each other in the same angular sector of the lumen perimeter, with or without malapposition; and/or 2) isolated struts located more or less at the center of the vessel without obvious connection to the expected adjacent strut pattern.
Scaffold pattern irregularities - Cohort B | 24 months
  Scaffold pattern irregularities are defined when struts are found in locations incongruent with the scaffold pattern, this is measured post-scaffold deployment and at follow up. They are classified into 2 categories: 1) 2 struts overhanging each other in the same angular sector of the lumen perimeter, with or without malapposition; and/or 2) isolated struts located more or less at the center of the vessel without obvious connection to the expected adjacent strut pattern.
Scaffold pattern irregularities - Cohort C | 36 months
  Scaffold pattern irregularities are defined when struts are found in locations incongruent with the scaffold pattern, this is measured post-scaffold deployment and at follow up. They are classified into 2 categories: 1) 2 struts overhanging each other in the same angular sector of the lumen perimeter, with or without malapposition; and/or 2) isolated struts located more or less at the center of the vessel without obvious connection to the expected adjacent strut pattern.

OTHER OUTCOMES:
Quantitative Coronary Angiography (QCA) derived parameters - All cohorts | Baseline
  Proximal 5mm side branch % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  Proximal 5mm side branch % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  Proximal 5mm side branch % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  Proximal 5mm side branch % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  In-segment Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  In-segment Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  In-segment Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  Proximal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  Proximal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  Proximal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  Distal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  Distal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  Distal Late Loss (LL) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - All cohorts | Baseline
  In-scaffold/in-stent, in-segment, proximal and distal Minimal Lumen Diameter (MLD) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  In-scaffold/in-stent, in-segment, proximal and distal Minimal Lumen Diameter (MLD) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  In-scaffold/in-stent, in-segment, proximal and distal Minimal Lumen Diameter (MLD) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  In-scaffold/in-stent, in-segment, proximal and distal Minimal Lumen Diameter (MLD) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - All cohorts | Baseline
  In-scaffold/in-stent, in-segment, proximal and distal % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  In-scaffold/in-stent, in-segment, proximal and distal % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  In-scaffold/in-stent, in-segment, proximal and distal % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  In-scaffold/in-stent, in-segment, proximal and distal % diameter stenosis (DS) postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort A | 12 months
  In-scaffold/in-stent, in-segment, proximal and distal angiographic binary restenosis rate postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 24 months
  In-scaffold/in-stent, in-segment, proximal and distal angiographic binary restenosis rate postnitrate
Quantitative Coronary Angiography (QCA) derived parameters - Cohort C | 36 months
  In-scaffold/in-stent, in-segment, proximal and distal angiographic binary restenosis rate postnitrate

CONTACTS AND LOCATIONS:
Overall Officials: Joanna J Wykrzykowska, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands